CLINICAL TRIAL: NCT03906422
Title: Comparison of Patient-reported Pain After Initial Archwire Placement With Three Types of Nickel-titanium Archwires: a Prospective Triple-blind, Randomized Controlled Clinical Trial
Brief Title: Comparison of Patient-reported Pain After Initial Archwire Placement
Acronym: Archwires
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18-1737
Record Dates: First submitted 2019-03-19; First posted 2019-04-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Orthodontic Discomfort; Pain, Orofacial
Keywords: Orthodontic; Pain
MeSH Terms: conditions — Facial Pain; Pain

STUDY DESIGN:
Intervention Model Description: prospective, triple-blind, randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator will assemble the opaque, sealed envelopes containing the archwires. The envelopes will be labeled "A", "B" or "C" corresponding to 0.016" Nitinol (3M Unitek, Monrovia, CA), 0.016" 27o CuNiTi (Ormco, Glendora, CA) or 0.016" 35o CuNiTi (Ormco, Glendora, CA) respectively. Randomization sequences will be created by using Research Randomizer online software. The investigator will enroll patients into the study. This trial will be completed with two blocks of 63 subjects each, one block per year, with subject randomization within each block.
  An independent third party will maintain possession of all envelopes and distribute as needed once a subject is enrolled and ready to receive fixed orthodontic appliances. The same independent third party will maintain a log with subject identification and consent forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- A: 0.016" Nitinol (Experimental): 0.016" Nitinol (3M Unitek, Monrovia, CA) archwire to be tied to the fixed orthodontic brackets at the initial bonding appointment.
  Interventions: Device: 3M Unitek 0.016 orthodontic archwire
- B: 0.016" Ormco 27oC NiTi (Experimental): 0.016" Ormco 27oC NiTi (Ormco, Glendora, CA) archwire to be tied to the fixed orthodontic brackets at the initial bonding appointment.
  Interventions: Device: Device: 0.016" Ormco 27oC NiTi orthodontic archwire
- C: 0.016" Ormco 35oC NiTi (Experimental): 0.016" Ormco 35oC NiTi (Ormco, Glendora, CA) archwire to be tied to the fixed orthodontic brackets at the initial bonding appointment.
  Interventions: Device: Device: 0.016" Ormco 35oC NiTi orthodontic archwire

INTERVENTIONS:
Device: 3M Unitek 0.016 orthodontic archwire — Placement of 3M Unitek 0.016 archwire for orthodontic treatment
  Arms: A: 0.016" Nitinol
Device: Device: 0.016" Ormco 27oC NiTi orthodontic archwire — Placement of 0.016" Ormco 27oC NiTi orthodontic archwire
  Arms: B: 0.016" Ormco 27oC NiTi
Device: Device: 0.016" Ormco 35oC NiTi orthodontic archwire — Placement of 0.016" Ormco 35oC NiTi orthodontic archwire
  Arms: C: 0.016" Ormco 35oC NiTi

SUMMARY:
Three different types of 'archwires' can be used in Orthodontic treatment, wire choice is decided by treating Orthodontist based on professional preference since research shows that all types are equally effective.

It is possible that one type of wire engenders more patient discomfort. This study will compare the discomfort levels engendered by the three wire types to determine if there is one that induces the least amount.

DETAILED DESCRIPTION:
Orthodontic treatment with fixed appliances has the potential to induce pain in patients. At the beginning of treatment, the orthodontist must determine which initial orthodontic archwire to insert. Among the more popular choices for initial leveling and aligning of the dental arches are small-sized, round-diameter nickel-titanium archwires. Various types of nickel-titanium (NiTi) archwires exist including stabilized martensitic wires (ie classic Nitinol), active austenitic wires (superelastic NiTi) and active martensitic wires (thermoelastic NiTi). The efficacy of these wire types has been heavily researched with no significant differences in the alignment timing of the dentition (treatment time to reach the final archwire). Pain differences from these wires has been inconclusive from conflicting past studies. It is of critical importance to determine whether one or more of these archwires leads to more discomfort for the patient than the others.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, with no significant systemic diseases or complications or special needs
2. Requiring a minimum of 1 dental arch (first molar to first molar) labial fixed orthodontic appliance banded/bonded in 1 appointment
3. All banded/bonded teeth can be ligated to initial archwire (no severely displaced or blocked out teeth).
4. Any planned dental extractions that is part of the orthodontic treatment plan must be carried out at least 3 weeks prior to or after initial orthodontic appliance bonding.
5. Age 12 years or older

Exclusion Criteria:

1. Currently taking or recently taken sulfonamides, monoamine oxidase inhibitors, tricyclic antidepressants, or phenothiazines
2. Currently taking physician-prescribed medical marijuana for the management of pain or recreational marijuana during the trial period
3. Metal-type (Nickel) allergies
4. Less than 12 years old
5. Same day use of analgesics prior to bonding
6. Treatment requiring dental extractions prior to or immediately after bonding of fixed appliance

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain score via Visual Analogue Score | 1 hour, 4 hour, 24 hour, 4 day and 7 day
  The primary outcome is the change in pain experienced by the study participant over the first week of therapy after insertion of the archwire.
  Pain is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of pain being experienced. The left end of the line is no pain where the right end is maximum (unimaginable) pain. The specific pain indicated is in the number of millimeters from the left end of the line. This is called the Visual Analogue Score (VAS) where the higher the number the more intense the pain.
  The difference in VAS pain scores from the initial VAS after archwire insertion (1 hour) to each measurement time (4 hour, 24 hour, 4 day and 7 day) over 7 days will indicate the change pain experience for each study participant.
  For each time point the mean and standard deviation of the change in VAS pain scores for the experimental groups will be calculated and compared for statistically significant differences.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado School of Dental Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The COMIRB approval and the consent forms specify that we cannot share PHI except as mandated by law. Therefore we do not intend to share any IPD to other researchers.

REFERENCES:
- [Background] Cioffi I, Piccolo A, Tagliaferri R, Paduano S, Galeotti A, Martina R. Pain perception following first orthodontic archwire placement--thermoelastic vs superelastic alloys: a randomized controlled trial. Quintessence Int. 2012 Jan;43(1):61-9. PMID 22259810
- [Background] Graf M, Alhammouri Q, Vieregge C, Lorenz B. The Bruckner transillumination test: limited detection of small-angle esotropia. Ophthalmology. 2011 Dec;118(12):2504-9. doi: 10.1016/j.ophtha.2011.05.016. PMID 21856007
- [Background] Krishnan V. Orthodontic pain: from causes to management--a review. Eur J Orthod. 2007 Apr;29(2):170-9. doi: 10.1093/ejo/cjl081. PMID 17488999
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093